CLINICAL TRIAL: NCT02478099
Title: MPDL3280A Treatment in Patients With Locally Advanced or Metastatic Solid Tumors After or During Investigational Imaging
Brief Title: MPDL3280A-treatment-IST-UMCG
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29755
Record Dates: First submitted 2015-05-21; First posted 2015-06-23 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: MPDL3280A; solid tumors
MeSH Terms: interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 Treatment with MPDL3280A (Experimental): Treatment with MPDL3280A
  Interventions: Drug: MPDL3280A

INTERVENTIONS:
Drug: MPDL3280A — Anti-PD-L1 antibody

SUMMARY:
To be able to evaluate the investigational imaging - 89Zr-MPDL3280A-PET, 89Zr-CD8 imaging and 18F-FB-IL2-PET - as complementary tools for selection of patients to be treated with MPDL3280A, within this treatment trial the investigators will assess safety, tolerability and anti-tumor activity of MPDL3280A in cancer patients, who have undergone investigational imaging.

DETAILED DESCRIPTION:
Encouraging clinical data emerging in the field of tumor immunotherapy have demonstrated that therapies focused on enhancing T cell responses against cancer can result in a significant survival benefit in patients with Stage IV cancer. PD-L1 is an extracellular protein that downregulates immune responses primarily in peripheral tissues through binding to its two receptors PD-1 and B7-1. Interruption of the PD L1/PD-1 pathway by the PD-L1 targeting antibody MPDL3280A, represents an attractive strategy to reinvigorate tumor-specific T cell immunity. For PD1/PD-L1 pathway inhibition PD-L1 tumor surface expression was proposed as a potential biomarker. In early clinical trials, PD-L1 expression has been associated with response to PD1/PD-L1 inhibition. However, other clinical trials reported response to PD1/PD-L1 checkpoint inhibitors in a big patient groups who were PD-L1-negative assessed by a single biopsy. Another obstacle to using PD-L1 expression as predictive biomarker might be its potential heterogeneous expression and fast dynamics PD-L1 tumor expression and whole body distribution, as well as baseline activation status of the immune system are being assessed in three investigational imaging trials MPDL3280A-img-042015, 89Zr-CD8 imaging or IL2-img--UMCG-2015.

To be able to evaluate the investigational imaging - 89Zr-MPDL3280A-PET, 89Zr-CD8 imaging and 18F-FB-IL2-PET - as complementary tools for selection of patients to be treated with MPDL3280A, within this treatment trial we will assess safety, tolerability and anti-tumor activity of MPDL3280A in cancer patients, who have undergone investigational imaging. Acquired data could lead to improved, more patient friendly, more easily accessible and possibly less expensive procedures for patient selection. Subsequently, the efficacy of (combinations of) checkpoint inhibition could also be improved, thus preventing unnecessary toxicity and reducing health care costs.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented locally advanced or metastatic solid tumor, whom in the opinion of the investigator, based on available clinical data, may benefit from treatment with anti PD-L1 immunotherapy .
2. Participation within the 18F-IL2 imaging trial (IL2-img-UMCG-2015) or 89Zr-MPDL3280A antibody imaging trial (MPDL3280A-img-042015) or CD8 imaging trial (ZED88082-img-UMCG-2018) before participation in the MPDL3280A treatment trial.
3. Subject must have undergone a fresh tumor biopsy for PD-L1 assessment performed as part of one of the investigational imaging trials.
4. Subjects are eligible if disease progression during or following first-line chemotherapy or any subsequent treatment lines for locally advanced or metastatic solid tumor whom, in the opinion of the investigator, based on available clinical data, may benefit from treatment with anti PD-L1 immunotherapy .

   ● Additional criteria for cancer of the urinary tract:
   * Subjects with disease progression during or following platinum-based adjuvant/neoadjuvant chemotherapy are eligible if ≤ 12 months have elapsed between the last treatment administration and the date of recurrence.

     ● Additional criteria for NSCLC:
   * Subjects with disease progression during or following platinum-based adjuvant/neoadjuvant chemotherapy or concurrent chemoradiation for NSCLC are eligible if ≤ 6 months have elapsed between the last treatment administration and the date of recurrence.
   * Subjects with a known sensitizing mutation in the epidermal growth factor receptor (EGFR) gene must also have experienced disease progression (during or after treatment) or intolerance to treatment with erlotinib, gefitinib, or another EGFR tyrosine kinase inhibitor (TKI).
   * Subjects with a known Anaplastic Lymphoma Kinase (ALK) fusion oncogene must also have experienced disease progression (during or after treatment) or intolerance to treatment with crizotinib or another ALK inhibitor.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy ≥12 weeks.
7. Signed Informed Consent Form.
8. Ability to comply with protocol.
9. Age ≥18 years.
10. Measurable disease, as defined by standard RECIST v1.1. Previously irradiated lesions should not be counted as target lesions.
11. Adequate hematologic and end organ function, defined by the following laboratory results obtained within ≤28 days prior to the first full dose of MPDL3280A:

    * ANC ≥1500 cells/μL (without granulocyte colony-stimulating factor support within 2 weeks prior to Cycle 1, Day 1).
    * WBC counts >2500/μL.
    * Lymphocyte count ≥500/μL.
    * Platelet count ≥100,000/μL (without transfusion within 2 weeks prior to Cycle 1, Day 1).
    * Hemoglobin ≥9.0 g/dL. Subjects may be transfused or receive erythropoietic treatment to meet this criterion.
    * AST, ALT, and alkaline phosphatase ≤ 2.5× the upper limit of normal (ULN), with the following exceptions:

      * Subjects with documented liver metastases: AST and/or ALT ≤ 5 × ULN.
      * Subjects with documented liver or bone metastases: alkaline phosphatase ≤ 5 × ULN.
    * Serum bilirubin ≤ 1.5 × ULN. Subjects with known Gilbert disease who have serum bilirubin level ≤ 3 × ULN may be enrolled.
    * INR and aPTT ≤ 1.5 × ULN. This applies only to subjects who are not receiving therapeutic anticoagulation; subjects receiving therapeutic anticoagulation should be on a stable dose.
    * Creatinine clearance ≥ 30 mL/min
12. For female subjects of childbearing potential and male subjects with partners of childbearing potential, agreement (by subject and/or partner) to use a highly effective form(s) of contraception (i.e., one that results in a low failure rate [< 1% per year] when used consistently and correctly) and to continue its use for 6 months after the last dose of MPDL3280A.

Exclusion Criteria:

1. Any approved anti-cancer therapy, including chemotherapy or hormonal therapy within ≤21 days prior to the first full dose of MPDL3280A; the following exceptions are allowed:

   * Hormone-replacement therapy or oral contraceptives.
   * TKIs approved for treatment of NSCLC discontinued >7 days prior to the first full dose of MPDL3280A. The baseline scan must be obtained after discontinuation of prior TKIs.
2. Treatment with any other investigational agent, other than the investigational tracer 89Zr-MPDL3280A, 18F-FB-IL2 or 89Zr-CD8-imaging, or participation in another clinical trial with therapeutic intent within 28 days prior to the first full dose of MPDL3280A.
3. Unstable brain metastases.
4. Unstable leptomeningeal disease.
5. Uncontrolled tumor-related pain.

   * Subjects requiring pain medication must be on a stable regimen at study entry.
   * Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastases causing nerve impingement) should be treated prior to enrollment. Subjects should be recovered from the effects of radiation. There is no required minimum recovery period.
   * Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
6. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Subjects with indwelling catheters (e.g., PleurX) are allowed.
7. Uncontrolled hypercalcemia (> 1.5 mmol/L ionized calcium or calcium >12 mg/dL or corrected serum calcium >ULN) or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy or denosumab.
8. Subjects, who are receiving bisphosphonate therapy or denosumab specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible.A second malignancy within 5 years prior to Cycle 1 Day 1, with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent, ductal carcinoma in situ treated surgically with curative intent).
9. Pregnant and lactating women.
10. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
11. Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cell products or any component of the MPDL3280A formulation.
12. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

    * Subjects with a history of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.
    * Subjects with controlled Type I diabetes mellitus on a stable dose of insulin regimen may be eligible for this study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

      * Rash must cover less than 10% of body surface area (BSA).
      * Disease is well controlled at baseline and only requiring low potency topical steroids.
      * No acute exacerbation of underlying condition within the previous 12 months (not requiring PUVA [psoralen plus ultraviolet A radiation], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, high potency or oral steroids).
13. History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.

    * History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
14. Serum albumin < 2.5 g/dL.
15. Positive test for HIV.
16. Subjects with active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.

    * Subjects with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg) are eligible. HBV DNA test must be performed in these subjects prior to Cycle 1, Day 1.
    * Subjects positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
17. Active tuberculosis.
18. Severe infections within 4 weeks prior to the first full dose of MPDL3280A, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
19. Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1.
20. Received therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1.

    ● Subjects receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
21. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the previous 3 months, unstable arrhythmias, or unstable angina.

    ● Subjects with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction <50% must be on a stable medical regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist if appropriate.
22. Major surgical procedure other than for diagnosis within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study.
23. Prior allogeneic bone marrow transplantation or solid organ transplant.
24. Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study.

    ● Influenza vaccination should be given during influenza season only (example: approximately October to March in the Northern Hemisphere). Subjects must not receive live, attenuated influenza vaccine (e.g. FluMist®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study treatment of within 5 months after the last dose of MPDL3280A.
25. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications.
26. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-PD-1, and anti-PD-L1 therapeutic antibodies.

    ● Subjects who have had prior anti-CTLA-4 treatment may be enrolled, provided the following requirements are met:
    * Minimum of 6 weeks from the last dose of anti-CTLA-4
    * No history of severe immune related adverse effects from anti-CTLA-4 (CTCAE Grade 3 and 4)
27. Treatment with systemic immunostimulatory agents (including but not limited to IFNs, IL-2) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to the first full dose of MPDL3280A.
28. Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to Cycle 1, Day 1.

    * Subjects who have received acute, low-dose, systemic immunosuppressant medications (e.g. a one-time dose of dexamethasone for nausea) may be enrolled in the study after discussion with and approval by the sponsor.
    * The use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g. fludrocortisone) for subjects with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of efficacy of MPDL3280A after investigational imaging as measured by objective response rate | 2 years

SECONDARY OUTCOMES:
To evaluate progression free survival (PFS) according to standard RECIST v1.1 as assessed by the investigator. | 2 years
To evaluate duration of response (DOR) according to standard RECIST v1.1 as assessed by the investigator. | 2 years
To evaluate DOR according to modified RECIST as assessed by the investigator. | 2 years
To evaluate ORR according to modified RECIST as assessed by the investigator. | 2 years
To evaluate PFS according to modified RECIST as assessed by the investigator. | 2 years
To evaluate the safety/tolerability (by analysis of adverse events) of MPDL3280A. | 2 years
  Safety assessment through:
  * Incidence, nature and severity of adverse events, including protocol-defined events of special interest, graded according to NCI CTCAE4.0
  * Changes in laboratory test results, vital signs and physical findings.
To determine the number of patients with and patients without tumor tracer uptake with 89Zr-MPDL3280A,89Zr-CD8 antibody study and 18F-FB-IL2 (as assessed in the accessory imaging trials) who also demonstrate response to MPDL3280A therapy. | 2 years
To correlate PD-L1 biopsy results as assessed in the trials MPDL3280A-img-042015, 89Zr-CD8 antibody imaging and IL2-img-UMCG-2015 to response to MPDL3280A therapy. | 2 years
To evaluate the utility of biopsy at the time of apparent disease progression to distinguish apparent increases in tumor volume related to the immunomodulatory activity of MPDL3280A from true disease progression | 2 years
The fecal microbiome will be analysed in related to antitumor effect. Feces sampling will be performed before treatment and at cycle three. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth de Vries, Professor, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Bensch F, van der Veen EL, Lub-de Hooge MN, Jorritsma-Smit A, Boellaard R, Kok IC, Oosting SF, Schroder CP, Hiltermann TJN, van der Wekken AJ, Groen HJM, Kwee TC, Elias SG, Gietema JA, Bohorquez SS, de Crespigny A, Williams SP, Mancao C, Brouwers AH, Fine BM, de Vries EGE. 89Zr-atezolizumab imaging as a non-invasive approach to assess clinical response to PD-L1 blockade in cancer. Nat Med. 2018 Dec;24(12):1852-1858. doi: 10.1038/s41591-018-0255-8. Epub 2018 Nov 26. PMID 30478423